CLINICAL TRIAL: NCT02581618
Title: Effect of One Cycle Remote Ischemic Preconditioning on Myocardial Injury After Percutaneous Coronary Interventions in Patients With Stable Coronary Artery Disease
Brief Title: Remote Ischemic Preconditioning in Elective Percutaneous Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Mustafa Adem YILMAZTEPE, Assistant Professor Of Medicine, Trakya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Trakya-Kardiyo-2015-1
Record Dates: First submitted 2015-10-19; First posted 2015-10-21 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Myocardial Ischemia; Ischemic Reperfusion Injury
Keywords: ischemic preconditioning; myocardial injury; percutaneous coronary intervention
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study group (Experimental): Remote ischemic preconditioning arm
  Blood pressure cuff will be inflated up to 200 mmHg in the non-dominant arm for 5 minutes before guiding catheter engagement.
  Interventions: Other: remote ischemic preconditioning
- Control group (No Intervention): No intervention will be performed. Percutaneous coronary intervention will be performed without ischemic preconditioning.

INTERVENTIONS:
Other: remote ischemic preconditioning — Blood pressure cuff inflation up to 200mmHg in the non-dominant arm before guiding catheter engagement
  Arms: Study group

SUMMARY:
Myocardial injury occurs after percutaneous coronary intervention due to micro emboli, ischemia-reperfusion injury or side branch occlusion. 3 cycles of ischemic preconditioning has been shown to be useful in preventing myocardial injury but it is not suitable to perform it especially in ad hoc interventions. In this study the investigators aim is to show whether one cycle remote ischemic preconditioning will be enough to prevent myocardial injury during percutaneous coronary intervention.

DETAILED DESCRIPTION:
About in one third of elective percutaneous coronary interventions (PCI) troponin release occurs showing myocardial necrosis. And it has been shown that myocardial necrosis due to coronary interventions has also adverse effects on long term prognosis.

Beneficial effects of of ischemic preconditioning in elective PCI and in coronary artery bypass surgery has been shown in several studies. In most of the trials 3 cycles of ischemia was performed, but this is time consuming and it's not suitable to apply it, in ad-hoc interventions. The investigators found one study showing that one cycle will also be enough to prevent troponin elevation after elective PCI.

The investigators aim was also to show that one cycle preconditioning performed just before coronary intervention will also be useful in preventing myocardial necrosis due to elective PCI.

ELIGIBILITY:
Inclusion Criteria

* Patients with stable coronary artery disease, in whom percutaneous coronary intervention is planned after coronary angiography
* Patients with informed consent

Exclusion Criteria:

* Acute or chronic renal failure (Creatinin clearance <60ml/dk)
* Acute heart failure
* Presence of hemodynamic instability
* Left main interventions
* Acute Coronary Syndrome
* Patients in whom cuff inflation is contraindicated in upper extremities (fistula, lymphoedema etc)
* Patients using nicorandil, glibenclamide or trimetazidine
* Patients not accepting the study
* Presence of troponin elevation before intervention
* Presence or suspicion of pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2015-05; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
hs-Troponin elevation | after 16 hours

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa A YILMAZTEPE, MD, Principal Investigator — Trakya University School Of Medicine, Department Of Cardiology, Edirne, TURKEY
Locations (1):
- Trakya University School Of Medicine, Department Of Cardiology, Edirne, Turkey (Türkiye)

REFERENCES:
- [Result] Pei H, Wu Y, Wei Y, Yang Y, Teng S, Zhang H. Remote ischemic preconditioning reduces perioperative cardiac and renal events in patients undergoing elective coronary intervention: a meta-analysis of 11 randomized trials. PLoS One. 2014 Dec 31;9(12):e115500. doi: 10.1371/journal.pone.0115500. eCollection 2014. PMID 25551671
- [Result] Xu X, Zhou Y, Luo S, Zhang W, Zhao Y, Yu M, Ma Q, Gao F, Shen H, Zhang J. Effect of remote ischemic preconditioning in the elderly patients with coronary artery disease with diabetes mellitus undergoing elective drug-eluting stent implantation. Angiology. 2014 Sep;65(8):660-6. doi: 10.1177/0003319713507332. Epub 2013 Oct 24. PMID 24163121
- [Result] Davies WR, Brown AJ, Watson W, McCormick LM, West NE, Dutka DP, Hoole SP. Remote ischemic preconditioning improves outcome at 6 years after elective percutaneous coronary intervention: the CRISP stent trial long-term follow-up. Circ Cardiovasc Interv. 2013 Jun;6(3):246-51. doi: 10.1161/CIRCINTERVENTIONS.112.000184. Epub 2013 May 21. PMID 23696599
- [Result] Zografos TA, Katritsis GD, Tsiafoutis I, Bourboulis N, Katsivas A, Katritsis DG. Effect of one-cycle remote ischemic preconditioning to reduce myocardial injury during percutaneous coronary intervention. Am J Cardiol. 2014 Jun 15;113(12):2013-7. doi: 10.1016/j.amjcard.2014.03.043. Epub 2014 Apr 1. PMID 24793669